CLINICAL TRIAL: NCT01657448
Title: Phase III, Prospective, Multicenter, Single-blind, Randomized, Superiority to Evaluate the Efficacy and Safety of Methenamine Association 250mg + Methylthioninium Chloride 20 mg Compared to Phenazopyridine 100 mg in Symptomatic Control of Dysuria
Brief Title: Efficacy Study of Methenamine + Methylthioninium Chloride vs Phenazopyridine for the Symptomatic Control of Dysuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CYSEMS0112
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Dysuria
Keywords: Symptom of Dysuria
MeSH Terms: conditions — Dysuria | interventions — Methenamine; Methylene Blue; Phenazopyridine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methenamine, Methylthioninium (Experimental)
  Interventions: Drug: Methenamine and Methylthioninium chloride
- Phenazopyridine (Active Comparator)
  Interventions: Drug: Phenazopyridine

INTERVENTIONS:
Drug: Methenamine and Methylthioninium chloride — • Ingesting two (02) tablets of the drug with a glass of water, every 8 hours for 3 days
  Arms: Methenamine, Methylthioninium
Drug: Phenazopyridine — • Ingesting two (02) tablets of the drug with a glass of water, every 8 hours for 3 days
  Other Names: Pyridium
  Arms: Phenazopyridine

SUMMARY:
The purpose of this study is to evaluate the efficacy of the combination of Methenamine + Methylthioninium chloride compared to phenazopyridine (comparator product) in the symptomatic relief of dysuria.

DETAILED DESCRIPTION:
* Single blind, randomized, prospective study.
* Length of experience: 03 days to 07 days.
* 03 visits (days 1, 4 and 7).
* Evaluation of the efficacy and safety of the medication.
* Shall be assessed for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate by agreeing to the terms proposed in the Clinical trial;
* Patients aged over 18 years of any ethnicity;
* Presence of dysuria with marking greater than or equal to 5 measured points on the categorical scale pre-treatment for pain symptom;

Exclusion Criteria:

* Patients who are febrile (axillary T º: ≥ 38 ° C), with back pain or lumbar;
* Patients with complicated clinical presentation of urinary tract infection;
* Patients with a history of allergy or intolerance to any known or suspected one of the ingredients of the product under investigation;
* Patients who are pregnant or during lactation, or childbearing potential and are not making use of effective contraception;
* Patients presenting with renal disease or severe liver disease, according to medical history and / or laboratory;
* Patients presenting with severe systemic disease according to the known medical history;
* Patients who received antibiotic treatment, anthelmintic within 7 days prior to study entry;
* Patients unable to understand the guidelines specified in this protocol or can not attend all study visits or unable to complete the log;
* Pregnancy or risk of pregnancy and lactating patients;
* Any finding of clinical observation (history and physical examination) that is interpreted by the physician investigator as a risk to the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in the symptomatic relief of dysuria | 3 days

SECONDARY OUTCOMES:
Safety of the study medication | 7 days
  To assess the safety of the study medication on the occurrence, type, intensity and frequency of adverse reactions during the treatment period.

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Centro de Medicina Reprodutiva Carlos Isaia Filho Ltda, Porto Alegre, Rio Grande do Sul
  - Marcio Antonio Pereira Clinica de Endocrinologia, São José dos Campos, São Paulo
  - AFIP, São Paulo
  - Savmed Clinica Médica S/C Ltda., São Paulo